CLINICAL TRIAL: NCT05175040
Title: PROphylactic Manual RotatIon in the Second stagE of Labor (PROMISE): a Randomized Controlled Trial
Brief Title: PROphylactic Manual RotatIon in the Second stagE of Labor
Acronym: PROMISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical challenges impeding enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Fisher, Assistant Professor of Obstetrics and Gynecology (Maternal Fetal Medicine), Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00215006
Record Dates: First submitted 2021-11-08; First posted 2022-01-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Labor Complication; Pregnancy Related
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both the study participant and her primary obstetrician will be blinded to the assigned randomization arm prior to delivery, as involvement in this research study should not change their care. Clinical management will be left to the discretion of each participant's primary obstetrician managing her labor, according to standard obstetrical care, who again will not be involved in the research-related study procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic manual rotation (Experimental): Prophylactic manual rotation involves a vaginal examination performed with an obstetric provider's hands to turn the baby from a position in which the baby's face is looking up in the direction of the ceiling (occiput posterior) or to the side (occiput transverse) to a position in which the baby's face is looking down in the direction of the mother's spine (occiput anterior). Prophylactic manual rotation will occur at the initiation of pushing once the individual achieves complete cervical dilation.
  Interventions: Procedure: Prophylactic manual rotation
- Sham rotation (Sham Comparator): Sham rotation involves a vaginal exam that obstetric providers commonly do with their hands to assess cervical dilation and fetal position during routine labor, and will occur at the initiation of pushing once the individual achieves complete cervical dilation.
  Interventions: Procedure: Sham rotation

INTERVENTIONS:
Procedure: Prophylactic manual rotation — Prophylactic manual rotation, performed in the experimental arm, involves a vaginal examination performed with an obstetric provider's hands to turn the baby from a position in which the baby's face is looking up in the direction of the ceiling (occiput posterior) or to the side (occiput transverse) to a position in which the baby's face is looking down in the direction of the mother's spine (occiput anterior). Prophylactic manual rotation will occur at the initiation of pushing once the individual achieves complete cervical dilation, performed by a trained study investigator (M.D. or midwife) to maintain blinding of the patient's primary obstetrician.
  Arms: Prophylactic manual rotation
Procedure: Sham rotation — Sham rotation, performed in the comparator arm, involves a vaginal exam that obstetric providers commonly do with their hands to assess cervical dilation and fetal position during routine labor, and will occur at the initiation of pushing once the individual achieves complete cervical dilation. Duration of the vaginal exam for sham rotation will be consistent with that used for prophylactic manual rotation and will be performed by a trained study investigator (M.D. or midwife) to maintain blinding of the patient's primary obstetrician.
  Arms: Sham rotation

SUMMARY:
This is a randomized controlled trial to determine whether prophylactic manual rotation for fetuses identified to have persistent occiput posterior or occiput transverse presentation (POP/OTP) at the initiation of the second stage of labor in nulliparous individuals reduces rates of operative delivery, second stage of labor duration, and resultant adverse clinical outcomes compared to standard management of the second stage of labor.

DETAILED DESCRIPTION:
This is a randomized controlled trial in which nulliparous individuals with a term, singleton gestation who undergo a trial of labor with neuraxial anesthesia and have a fetus presenting with persistent occiput posterior or occiput transverse presentation (POP/OTP) confirmed by ultrasound at the initiation of the second stage of labor will be randomized to either prophylactic manual rotation or sham rotation. The study aims to evaluate whether prophylactic manual rotation reduces the incidence of operative delivery (a composite of cesarean and operative vaginal delivery), second stage of labor duration, and maternal and neonatal morbidity among nulliparous individuals with a fetus with POP/OTP at the initiation of the second stage of labor.

Individuals will be screened for eligibility upon admission to Labor and Delivery and approached for potential recruitment with informed consent obtained on enrollment. Once women achieve complete cervical dilation and within the first fifteen minutes of commencement of pushing, a bedside ultrasound will be performed to determine the fetal position. Those with POP/OTP will be randomized at that time point to either prophylactic manual rotation or sham rotation. The patient's primary obstetrician will be blinded to the randomization arm. The electronic health record will be reviewed and used to assess trial outcomes. The study will enroll 350 individuals, powered to detect a 15% reduction in operative delivery (instrumental vaginal delivery or cesarean section) with prophylactic manual rotation of POP/OTP, from a baseline risk of 50% without manual rotation to 35% with prophylactic rotation at initiation of the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Age 18 years or greater
* English-speaking
* Nulliparous
* Singleton gestation
* Planning a vaginal birth
* Have neuraxial anesthesia
* Term gestation (≥37 weeks' gestation)
* Ruptured membranes
* Complete cervical dilation
* Cephalic presenting fetus
* Fetus presenting with occiput posterior or occiput transverse position confirmed by ultrasound

Exclusion Criteria:

* Pregnancies with intrauterine fetal demise
* Pregnancies affected by major fetal anomaly
* Maternal or fetal contraindication to vaginal delivery, including operative vaginal delivery
* Fetal malpresentation, including brow or face presentation
* Category III fetal heart rate tracing at time of randomization
* Duration of pushing already exceeding 15 minutes in the second stage of labor
* Lack of other inclusion criteria as described above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants in each group who undergo operative delivery | From randomization until delivery, up to 5 hours
  Number of participants in each group who undergo a cesarean section or an instrumental delivery (vacuum or forceps) as a composite outcome

SECONDARY OUTCOMES:
Number of participants in each group who undergo operative vaginal delivery | From randomization until delivery, up to 5 hours
  Number of participants in each group who undergo an instrumental vaginal delivery with vacuum or forceps
Number of participants in each group who undergo cesarean delivery | From randomization until delivery, up to 5 hours
  Number of participants in each group who undergo a cesarean section
Number of minutes in the second stage of labor in each group | From randomization until delivery, up to 300 minutes
  Number of minutes participants in each group spend in the second stage of labor
Number of participants in each group with composite maternal morbidity | From randomization until hospital discharge, an expected average of 3 days
  Number of participants in each group with a composite of the following individual adverse maternal outcomes: obstetric anal sphincter injury (i.e. 3rd or 4th degree perineal lacerations), postpartum hemorrhage (i.e. estimated blood loss as defined by >1000ml), blood product transfusion, intrapartum chorioamnionitis diagnosed in the second stage of labor, or postpartum endometritis
Number of participants in each group with maternal intrapartum chorioamnionitis diagnosed in the second stage of labor | From randomization until delivery, up to 5 hours
  Number of participants in each group who are diagnosed with intrapartum chorioamnionitis during the second stage of labor as defined by fever greater than 100.4 Fahrenheit in the intrapartum period and at least one additional clinical factor (fundal tenderness, maternal tachycardia, fetal tachycardia, or purulent discharge) with initiation of a therapeutic antibiotic regimen in the second stage of labor
Number of participants in each group with postpartum endometritis | From delivery until hospital discharge, an expected average of 3 days
  Number of participants in each group who experience postpartum endometritis as defined by fever greater than 100.4 Fahrenheit and one additional clinical factor (fundal tenderness or purulent lochia) in the postpartum period with the initiation of a therapeutic antibiotic regimen in the postpartum period
Number of participants in each group with postpartum hemorrhage | From randomization until hospital discharge, an expected average of 3 days
  Number of participants in each group with postpartum hemorrhage (i.e. estimated blood loss as defined by >1000ml)
Number of participants in each group who require blood product transfusion | From randomization until hospital discharge, an expected average of 3 days
  Number of participants in each group who require blood product transfusion
Number of participants in each group who experience obstetric anal sphincter injury (i.e. a composite of 3rd or 4th degree perineal lacerations) | From randomization until delivery, up to 5 hours
  Number of participants in each group with 3rd or 4th degree perineal lacerations as a composite outcome
Number of participants in each group with composite severe neonatal morbidity | From delivery until hospital discharge, up to 28 days of life
  Number of participants in each group with neonates with the composite of the following individual adverse neonatal outcomes: 5-minute Apgar score <5, arterial cord pH ≤7.00 or base excess ≤-12 milliequivalents/L, shoulder dystocia, hypoxic-ischemic encephalopathy requiring hypothermic therapy or neonatal subgaleal or intracranial hemorrhage, neonatal intensive care unit (NICU) admission, or neonatal sepsis
Number of participants in each group who experience neonatal death | From delivery until hospital discharge, up to 28 days of life
  Number of participants in each group with neonates who experience neonatal death after delivery prior to hospital discharge
Number of participants in each group affected by neonatal intensive care unit (NICU) admission | From delivery until hospital discharge, up to 28 days of life
  Number of participants in each group with a neonate that requires neonatal intensive care unit (NICU) admission following delivery
Number of days a participant in each group has a neonate requiring neonatal intensive care unit (NICU) admission | From delivery until hospital discharge, up to 28 days of life
  Number of days a participant in each group has a neonate that is admitted to the neonatal intensive care unit (NICU) following delivery
Number of participants in each group with a neonate with neonatal 5-minute Apgar score <5 | From delivery up to 5 minutes of life
  Number of participants in each group with a neonate that has an Apgar score less than 5 at 5 minutes of life
Number of participants in each group with a neonate with neonatal umbilical arterial cord pH ≤7.00 or base excess ≤-12 milliequivalents/L | At time of delivery
  Number of participants in each group with a neonate that has an umbilical arterial cord pH less than or equal to 7.00 or base excess less than or equal to -12 milliequivalents/L as a composite outcome
Number of participants in each group who experiences intrapartum shoulder dystocia | From randomization until delivery, up to 5 hours
  Number of participants in each group that experiences a shoulder dystocia at delivery
Number of participants in each group with a neonate with neonatal hypoxic-ischemic encephalopathy requiring hypothermic therapy or neonatal subgaleal or intracranial hemorrhage | From delivery until hospital discharge, up to 28 days of life
  Number of participants in each group with a neonate that experiences development of hypoxic-ischemic encephalopathy requiring hypothermic therapy or development of subgaleal or intracranial hemorrhage as a result of birth trauma or other delivery event
Number of participants in each group with a neonate with neonatal sepsis | From delivery until hospital discharge, up to 28 days of life
  Number of participants in each group with a neonate that experiences neonatal sepsis as defined by pathogenic bacterial infection confirmed in blood or cerebrospinal fluid culture

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Fisher, MD MPH, Study Director — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Morton R, Burton AE, Kumar P, Hyett JA, Phipps H, McGeechan K, de Vries BS. Cesarean delivery: Trend in indications over three decades within a major city hospital network. Acta Obstet Gynecol Scand. 2020 Jul;99(7):909-916. doi: 10.1111/aogs.13816. Epub 2020 Feb 12. PMID 31976544
- [Background] Operative Vaginal Birth: ACOG Practice Bulletin, Number 219. Obstet Gynecol. 2020 Apr;135(4):e149-e159. doi: 10.1097/AOG.0000000000003764. PMID 32217976
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 165: Prevention and Management of Obstetric Lacerations at Vaginal Delivery. Obstet Gynecol. 2016 Jul;128(1):e1-e15. doi: 10.1097/AOG.0000000000001523. PMID 27333357
- [Background] Senecal J, Xiong X, Fraser WD; Pushing Early Or Pushing Late with Epidural study group. Effect of fetal position on second-stage duration and labor outcome. Obstet Gynecol. 2005 Apr;105(4):763-72. doi: 10.1097/01.AOG.0000154889.47063.84. PMID 15802403
- [Background] Lieberman E, Davidson K, Lee-Parritz A, Shearer E. Changes in fetal position during labor and their association with epidural analgesia. Obstet Gynecol. 2005 May;105(5 Pt 1):974-82. doi: 10.1097/01.AOG.0000158861.43593.49. PMID 15863533
- [Background] Fitzpatrick M, McQuillan K, O'Herlihy C. Influence of persistent occiput posterior position on delivery outcome. Obstet Gynecol. 2001 Dec;98(6):1027-31. doi: 10.1016/s0029-7844(01)01600-3. PMID 11755548
- [Background] Ponkey SE, Cohen AP, Heffner LJ, Lieberman E. Persistent fetal occiput posterior position: obstetric outcomes. Obstet Gynecol. 2003 May;101(5 Pt 1):915-20. doi: 10.1016/s0029-7844(03)00068-1. PMID 12738150
- [Background] Macara LM, Murphy KW. The contribution of dystocia to the cesarean section rate. Am J Obstet Gynecol. 1994 Jul;171(1):71-7. doi: 10.1016/s0002-9378(94)70080-x. PMID 7794300
- [Background] Le Ray C, Serres P, Schmitz T, Cabrol D, Goffinet F. Manual rotation in occiput posterior or transverse positions: risk factors and consequences on the cesarean delivery rate. Obstet Gynecol. 2007 Oct;110(4):873-9. doi: 10.1097/01.AOG.0000281666.04924.be. PMID 17906022
- [Background] Carseldine WJ, Phipps H, Zawada SF, Campbell NT, Ludlow JP, Krishnan SY, De Vries BS. Does occiput posterior position in the second stage of labour increase the operative delivery rate? Aust N Z J Obstet Gynaecol. 2013 Jun;53(3):265-70. doi: 10.1111/ajo.12041. Epub 2013 Jan 24. PMID 23346873
- [Background] Benavides L, Wu JM, Hundley AF, Ivester TS, Visco AG. The impact of occiput posterior fetal head position on the risk of anal sphincter injury in forceps-assisted vaginal deliveries. Am J Obstet Gynecol. 2005 May;192(5):1702-6. doi: 10.1016/j.ajog.2004.11.047. PMID 15902181
- [Background] Wu JM, Williams KS, Hundley AF, Connolly A, Visco AG. Occiput posterior fetal head position increases the risk of anal sphincter injury in vacuum-assisted deliveries. Am J Obstet Gynecol. 2005 Aug;193(2):525-8; discussion 528-9. doi: 10.1016/j.ajog.2005.03.059. PMID 16098883
- [Background] Cheng YW, Shaffer BL, Caughey AB. Associated factors and outcomes of persistent occiput posterior position: A retrospective cohort study from 1976 to 2001. J Matern Fetal Neonatal Med. 2006 Sep;19(9):563-8. doi: 10.1080/14767050600682487. PMID 16966125
- [Background] Cheng YW, Shaffer BL, Caughey AB. The association between persistent occiput posterior position and neonatal outcomes. Obstet Gynecol. 2006 Apr;107(4):837-44. doi: 10.1097/01.AOG.0000206217.07883.a2. PMID 16582120
- [Background] Le Ray C, Deneux-Tharaux C, Khireddine I, Dreyfus M, Vardon D, Goffinet F. Manual rotation to decrease operative delivery in posterior or transverse positions. Obstet Gynecol. 2013 Sep;122(3):634-40. doi: 10.1097/AOG.0b013e3182a10e43. PMID 23921875
- [Background] Shaffer BL, Cheng YW, Vargas JE, Caughey AB. Manual rotation to reduce caesarean delivery in persistent occiput posterior or transverse position. J Matern Fetal Neonatal Med. 2011 Jan;24(1):65-72. doi: 10.3109/14767051003710276. Epub 2010 Mar 30. PMID 20350240
- [Background] Reichman O, Gdansky E, Latinsky B, Labi S, Samueloff A. Digital rotation from occipito-posterior to occipito-anterior decreases the need for cesarean section. Eur J Obstet Gynecol Reprod Biol. 2008 Jan;136(1):25-8. doi: 10.1016/j.ejogrb.2006.12.025. Epub 2007 Mar 21. PMID 17368909
- [Background] Graham K, Phipps H, Hyett JA, Ludlow JP, Mackie A, Marren A, De Vries B. Persistent occiput posterior: OUTcomes following digital rotation: a pilot randomised controlled trial. Aust N Z J Obstet Gynaecol. 2014 Jun;54(3):268-74. doi: 10.1111/ajo.12192. Epub 2014 Mar 16. PMID 24627988
- [Background] Phipps H, Hyett JA, Kuah S, Pardey J, Matthews G, Ludlow J, Narayan R, Santiagu S, Earl R, Wilkinson C, Bisits A, Carseldine W, Tooher J, McGeechan K, de Vries B. Persistent occiput posterior position outcomes following manual rotation: a randomized controlled trial. Am J Obstet Gynecol MFM. 2021 Mar;3(2):100306. doi: 10.1016/j.ajogmf.2021.100306. Epub 2021 Jan 6. PMID 33418103
- [Background] Broberg JC, Caughey AB. A randomized controlled trial of prophylactic early manual rotation of the occiput posterior fetus at the beginning of the second stage vs expectant management. Am J Obstet Gynecol MFM. 2021 Mar;3(2):100327. doi: 10.1016/j.ajogmf.2021.100327. Epub 2021 Feb 2. PMID 33545441
- [Background] Blanc J, Castel P, Mauviel F, Baumstarck K, Bretelle F, D'Ercole C, Haumonte JB. Prophylactic manual rotation of occiput posterior and transverse positions to decrease operative delivery: the PROPOP randomized clinical trial. Am J Obstet Gynecol. 2021 Oct;225(4):444.e1-444.e8. doi: 10.1016/j.ajog.2021.05.020. Epub 2021 May 24. PMID 34033811
- [Background] Le Ray C, Goffinet F. [Manual rotation of occiput posterior presentation]. Gynecol Obstet Fertil. 2011 Oct;39(10):575-8. doi: 10.1016/j.gyobfe.2011.08.038. Epub 2011 Sep 15. French. PMID 21924659
- [Background] Verhaeghe C, Parot-Schinkel E, Bouet PE, Madzou S, Biquard F, Gillard P, Descamps P, Legendre G. The impact of manual rotation of the occiput posterior position on spontaneous vaginal delivery rate: study protocol for a randomized clinical trial (RMOS). Trials. 2018 Feb 14;19(1):109. doi: 10.1186/s13063-018-2497-7. PMID 29444695
- [Background] Verhaeghe C, Corroenne R, Spiers A, Descamps P, Gascoin G, Bouet PE, Parot-Schinkel E, Legendre G. Delivery Mode After Manual Rotation of Occiput Posterior Fetal Positions: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):999-1006. doi: 10.1097/AOG.0000000000004386. PMID 33957650